CLINICAL TRIAL: NCT06476860
Title: Proteinuria During Sepsis and Septic Shock: Characterization and Association With Acute Respiratory Distress Syndrome
Brief Title: Proteinuria During Sepsis and Septic Shock: Characterization and Association With ARDS
Acronym: ALBUREA
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal André Grégoire (Other)
Responsible Party: Sponsor
Other Study IDs: GHT_CHIM RNI20221130
Record Dates: First submitted 2024-05-30; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-05

CONDITIONS: Sepsis and Septic Shock
Keywords: proteinuria; septic shock; sepsis; Acute Respiratory Distresse Syndrome
MeSH Terms: conditions — Sepsis; Shock, Septic; Proteinuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients suspected of sepsis or septic shock

SUMMARY:
ARDS is a pulmonary edema injury. Among its etiologies, it can be secondary to septic shock. Managing septic shock involves hemodynamic optimization with significant fluid and sodium inputs. Fluid and sodium inputs in ARDS worsen respiratory failure through capillary leakage, and a restrictive input strategy is clinically beneficial (reduced mechanical ventilation duration and ICU stay). Predicting ARDS onset in septic shock allows for optimized fluid and sodium input management, adopting a restrictive rather than liberal approach to minimize deterioration in respiratory function.

DETAILED DESCRIPTION:
Septic shock remains highly fatal, causing multi-organ failure including hemodynamic, pulmonary, neurological, renal, hematologic, and hepatic. These failures stem from generalized inflammatory aggression leading to endothelial dysfunction, especially at the capillary level. Pulmonary failure secondary to septic shock is characterized by edema, with ARDS being the most severe form. Sepsis is the second most common cause of ARDS after pneumonia. The incidence of ARDS in severe sepsis is about 6%, and its occurrence is an independent factor contributing to increased mortality.

These failures significantly impact the management of septic shock, where early and often agressive, vascular filling is standard for hemodynamic failure. Conversely, the onset of ARDS onset warrants limiting hydro-sodium inputs. Currently, there are no data predicting the occurrence of ARDS patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 and older admitted to the intensive care unit for suspected sepsis or septic shock.

Exclusion Criteria:

* Minors or opposition to participation.
* Chronic dialysis patients
* Organ transplant recipients
* Confirmed urinary tract infection
* Subject with macroscopic hematuria
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients suspected of sepsis or septic shock until 100 patients are enrolled. Infection diagnosis is based on systemic clinical signs (fever) or local inflammatory signs, biological evidence, and suspicion or confirmation of an infectious agent. The diagnosis of sepsis involves infection accompanied by organ failure, which may manifest as cardiovascular, respiratory, neurological, metabolic, renal, coagulation, or hepatic impairment. These signs may precede hypotension or occur without it.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of proteinuria in the first 24 hours (H0 and H24) of septic shock. | 24 hours
  relationship between proteinuria kinetics in the first 24 hours (H0 and H24) of septic shock and presence of ARDS at H72

SECONDARY OUTCOMES:
measurement of albuminuria urinary IgG at H0 and H24 | 24 hours
  Evaluation of the association between proteinuria kinetics and the onset of hemodynamic failure, renal failure, duration of mechanical ventilation, ICU stay, and hospital mortality
measurement of alpha-1-microglobulin at H0 and H24 | 24 hours
  Evaluation of the association between proteinuria kinetics and the onset of hemodynamic failure, renal failure, duration of mechanical ventilation, ICU stay, and hospital mortality
measurement of urinary IgG at H0 and H24 | 24 hours
  Evaluation of the association between proteinuria kinetics and the onset of hemodynamic failure, renal failure, duration of mechanical ventilation, ICU stay, and hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Andre Gregoire, Montreuil, France

REFERENCES:
- [Result] Iba T, Levy JH. Derangement of the endothelial glycocalyx in sepsis. J Thromb Haemost. 2019 Feb;17(2):283-294. doi: 10.1111/jth.14371. Epub 2019 Feb 3. PMID 30582882